CLINICAL TRIAL: NCT07119138
Title: The Effect of Emotional Freedom Technique on State Exam Anxiety Levels of Nursing Students: A Randomized Controlled Trial
Brief Title: Effect of Emotional Freedom Technique on Nursing Students Exam Anxiety
Acronym: EFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Mahsum KORKUTAN, Research assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25000
Record Dates: First submitted 2025-07-11; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Pre-Exam Anxiety; Emotional Freedom Technique
Keywords: Pre-Exam Anxiety; Nursing student; Mind-Body Therapies; Surgical nursing; Randomised controlled trial

STUDY DESIGN:
Intervention Model Description: It was planned to assign students who meet the selection criteria for the study and volunteer to participate in the study to the EFT group and the control group using the block randomization method. Blocks of 8 will be created according to the number of volunteer participants.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To prevent assignment bias in the study, blocks will be created by a statistician. The letters representing the experimental and control groups (A and B) will be determined by drawing lots. Because the researcher must have students administer the EFT one-on-one, blinding will not be possible during the application. After determining the students who meet the inclusion criteria and provide informed consent for assignment to groups (assignment blinding), researcher MK, who will be administering the EFT, will be notified by researcher SF. Students will not be informed of their group placement. After data collection, the groups will be coded as A and B in the dataset created by the researcher, and the codes will not be disclosed to the statistician conducting the analyses before reporting (blind technique).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): EFT arm
  Interventions: Behavioral: Emotional Freedom Technique
- Control (No Intervention): Control arm

INTERVENTIONS:
Behavioral: Emotional Freedom Technique — Emotional Freedom Technique (EFT) is used as an effective method for managing various adverse conditions, including the reduction of exam anxiety. Although there are several studies in the literature on this topic, research conducted specifically with nursing students remains limited. In particular, the Surgical Nursing course is a fundamental subject offered in the second year of nursing education, encompassing both theoretical and clinical components. Academic success in this course is an important indicator of the quality of nursing education. Therefore, as a surgical nursing instructor, it is believed that reducing exam anxiety can positively influence student performance.
  This study also aims to improve student success through anxiety management. To date, no studies addressing this issue with nursing students have been found in the literature.
  Arms: Experimental

SUMMARY:
Aim: This study was conducted to evaluate the effect of Emotional Freedom Technique (EFT) on the state exam anxiety levels of nursing students.

Background: Exam anxiety is a common problem among nursing students. EFT has emerged as a complementary method to reduce exam anxiety. However, experimental studies on this subject are limited in the literature.

Design: Randomized controlled trial design.

Methods: This study was carried out with second-year students enrolled in the Surgical Nursing course at the Faculty of Nursing of a state university. Participants were assigned to intervention and control groups using simple random sampling. One hour before the exam, all students were present in the exam hall. While the intervention group received EFT, the control group was given free time. Data were collected using the State Test Anxiety Scale (STAS) and the Subjective Units of Distress Scale (SUD). Descriptive statistics, normality tests (Shapiro-Wilk/Kolmogorov-Smirnov), independent and paired samples t-test, Mann-Whitney U test, Wilcoxon test, and two-way mixed ANOVA were used for data analysis. The significance level was set at p<0.05.

Outcomes: There were no significant differences between the groups in the pre-test STAS total and subscale scores or SUD scores. However, post-test results revealed statistically significant differences between the intervention and control groups in all measurements (p<0.05), with effect sizes ranging from medium to large. The time and group-time interaction effects for STAS total and subscale scores and SUD scores were also significant (p<0.05), and the effect size of the change over time was determined to be large (η² > 0.14).

Conclusion: This study demonstrated that EFT is effective in reducing exam anxiety among nursing students. EFT should be considered a complementary intervention in managing exam anxiety. It is recommended that EFT be integrated into the support services provided to students prior to examinations.

DETAILED DESCRIPTION:
Test anxiety is a set of phenomenological, physiological, and behavioral responses that accompany anxiety about possible negative outcomes or failure in an exam or assessment situation. Test anxiety is a form of situational anxiety and is an important factor affecting students' health and academic performance throughout their educational journey. It is stated in the literature that students' past experiences and beliefs, family attitudes, perceptions about course load, and time management skills can have an impact on test anxiety.

It is emphasized that low levels of anxiety support creativity and development in students, while high levels of anxiety can cause emotional and physiological arousal, leading to significant limiting behaviors such as excessive restlessness and anxiety.

It is stated that anxious students are easily distracted during exams and have difficulty understanding instructions. The severity of exam anxiety in students can reach clinical dimensions and negatively affect daily life, the educational process and career advancement . In the literature, it is stated that exam anxiety is associated with a number of negative variables such as increased risk of anxiety and depression in later life, difficulties in participating in teaching content, lack of attention, shorter concentration periods, decreased learning problems, low exam performance and decrease in academic achievement. Studies specifically link test anxiety to academic success and show that high test anxiety leads to a decrease in academic success. Nursing students also encounter various stressful situations throughout their academic journey.

Nursing education includes both theoretical and practical teaching processes, and this curriculum includes intense course loads, rigorous exams, and pressure to achieve a high GPA in a competitive environment. Clinical education, in which skill development is especially assessed, stands out as one of the first steps in acquiring professional skills and creates a significant source of stress and anxiety in nursing students, becoming a situation that needs to be managed. In the literature, it is stated that the test anxiety experienced by nursing students worldwide is one of the most important problems that prevent the acquisition of professional skills, and it is reported that 50% to 100% of nursing students experience test anxiety at least once during their undergraduate education. Therefore, there is a need for effective therapeutic interventions using complementary methods to reduce the negative effects of exam anxiety among nursing students. When the studies are examined, it is seen that many methods such as hand massage, music therapy, aromatherapy, auriculotherapy, gum chewing, trust training, coping program, animal-assisted intervention, guided imagery, expressive writing, mindfulness exercises, relaxation with cognitive behavioral methods are used to reduce exam anxietyç. It is known that another method used in the management of exam anxiety is the Emotional Freedom Technique (EFT).

EFT is an evidence-based therapeutic method that combines cognitive reframing and exposure therapies with light tapping on acupuncture points (acupressure) to induce relaxation. This method, which involves touching specific acupressure points while focusing on emotional concerns, stimulates the body's energy meridians to promote relaxation. EFT, which has a mechanism of action that alters emotional responses through limbic pathways by reactivating disturbing memories or triggers and allows the release of intense emotional experiences, is used to improve an individual's negative emotions and manage associated emotional and physical disorders. In the literature, EFT has been shown to be effective on depression, phobias, post-traumatic stress disorder, pain, insomnia, autoimmune diseases, professional performance, sports performance, anxiety, and exam anxiety. EFT studies on students show that this technique has a very therapeutic effect in overcoming anxiety and student motivation problems. Many other studies have also found that EFT significantly reduces exam anxiety in nursing students who receive clinical and theoretical training with an intensive curriculum.

As a self-help tool, EFT is easy to learn and apply, provides effective results in a short time and has been proven to reduce exam anxiety. EFT and exam anxiety have been studied limitedly internationally and two studies on this subject have been found at the national level. In this direction, this study aims to contribute to the literature by evaluating the effect of EFT on exam anxiety in nursing students. Surgical Diseases Nursing course is one of the basic courses given in the second year of nursing education, including theoretical and clinical components. The academic success of students in this course is decisive in terms of the quality of nursing education. Therefore, as a surgical nursing instructor, it is thought that reducing exam anxiety will positively affect student success. This study also aims to increase student success through anxiety management.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers to participate in the study • Qualified to take the final exam of the Surgical Diseases Nursing course

Exclusion Criteria:

* Refusing to participate in the study
* Receiving psychiatric treatment/receiving psychological support
* Failing the Surgical Diseases Nursing course application

Removal criteria

* A student who did not take the course exam due to illness, delay, or similar reasons
* Someone who wishes to withdraw from the study during the implementation phase after having agreed to participate.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Exam Anxiety Scale scores | The intervention started one hour before the surgical nursing final exam. The STAS pre-test was administered one hour before the exam, followed by the intervention (EFT). After the intervention, the STAS post-test was conducted.
  Change in Exam Anxiety Scale (STAS) scores before and after the intervention

SECONDARY OUTCOMES:
Change in Subjective Units of Distress (SUD) scores | The intervention started one hour before the surgical nursing final exam. The SUD pre-test was administered one hour before the exam, followed by the intervention (EFT). After the intervention, the SUD post-test was conducted
  Change in Subjective Units of Distress (SUD) scores before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Faculty of Theology, Laboratory, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participants' personal information will not be shared. Demographic data and scale scores included in the statistical analysis are being considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years from the article publication
Access Criteria: In case of a request for research purposes, the researcher will be directed to the drive link provided by SF.

REFERENCES:
- [Background] Bach D, Groesbeck G, Stapleton P, Sims R, Blickheuser K, Church D. Clinical EFT (Emotional Freedom Techniques) Improves Multiple Physiological Markers of Health. J Evid Based Integr Med. 2019 Jan-Dec;24:2515690X18823691. doi: 10.1177/2515690X18823691. PMID 30777453
- [Background] Boath, E., Stewart, A., & Carryer, A. (2013). Tapping for success: A pilot study to explore if emotional freedom techniques (EFT) can reduce anxiety and enhance academic performance in university students. Innovative Practice in Higher Education, 1(3).
- [Background] Church, D. (2013). The EFT manual. Hay House, Inc.
- [Background] Church D, Stapleton P, Vasudevan A, O'Keefe T. Clinical EFT as an evidence-based practice for the treatment of psychological and physiological conditions: A systematic review. Front Psychol. 2022 Nov 10;13:951451. doi: 10.3389/fpsyg.2022.951451. eCollection 2022. PMID 36438382
- [Background] Cici R, Ozkan M. Effects on Anxiety and Vital Signs of the Emotional Freedom Technique and Music Before Surgery for Lumbar Disc Hernia. Altern Ther Health Med. 2022 Jul;28(5):20-27. PMID 34097649
- [Background] Clond M. Emotional Freedom Techniques for Anxiety: A Systematic Review With Meta-analysis. J Nerv Ment Dis. 2016 May;204(5):388-95. doi: 10.1097/NMD.0000000000000483. PMID 26894319
- [Background] Craig G. (2011). The EFT manual (2nd ed.). Fulton, CA: Energy Psychology Press.
- [Background] Craig, G., & Fowlie, A. (1995). Emotional freedom techniques. Self-published manual. The Sea Ranch.
- [Background] Dincer B, Inangil D. The effect of Emotional Freedom Techniques on nurses' stress, anxiety, and burnout levels during the COVID-19 pandemic: A randomized controlled trial. Explore (NY). 2021 Mar-Apr;17(2):109-114. doi: 10.1016/j.explore.2020.11.012. Epub 2020 Dec 3. PMID 33293201
- [Background] Dincer B, Ozcelik SK, Ozer Z, Bahcecik N. Breathing therapy and emotional freedom techniques on public speaking anxiety in Turkish nursing students: A randomized controlled study. Explore (NY). 2022 Mar-Apr;18(2):226-233. doi: 10.1016/j.explore.2020.11.006. Epub 2020 Dec 2. PMID 33309466
- [Background] Efroliza, E. (2023). The Effect of Mentoring and Emotional Freedom Technique (M-EFT) on Nurses Students' Readiness and Anxiety Facing Competency Tests. Indonesıan Nursıng Journal of Educatıon And Clınıc (Injec), 8(1), 22-30
- [Background] Azzizadeh Forouzi M, Taebi M, Samarehfekri A, Rashidipour N. The effect of emotional freedom techniques on test anxiety in Iranian Paramedical students: a randomized controlled trial study. Ann Med Surg (Lond). 2024 Apr 3;86(5):2745-2751. doi: 10.1097/MS9.0000000000002023. eCollection 2024 May. PMID 38694321
- [Background] Guler, S., Demir, G., & Sahan, S. (2023). The effect of aromatherapy performed to nursing students on the level of test-taking anxiety and academic achievement. International Journal of Caring Sciences, 16(3), 1728.
- [Background] Hendricks-Patel S, Harvey K. Emotional Freedom Technique for Stress Reduction in Nursing Students: A Pilot Project. J Nurs Educ. 2025 Jul;64(7):436-439. doi: 10.3928/01484834-20250108-03. Epub 2025 Mar 13. PMID 40071786
- [Background] Huntley CD, Young B, Temple J, Longworth M, Smith CT, Jha V, Fisher PL. The efficacy of interventions for test-anxious university students: A meta-analysis of randomized controlled trials. J Anxiety Disord. 2019 Apr;63:36-50. doi: 10.1016/j.janxdis.2019.01.007. Epub 2019 Feb 6. PMID 30826687
- [Background] İnangil, D., Vural, P. I., Doğan, S., & Körpe, G. (2020). Effectiveness of music therapy and emotional freedom technique on test anxiety in Turkish nursing students: a randomised controlled trial. European Journal of Integrative Medicine, 33, 101041.
- [Background] Kalroozi F, Moradi M, Ghaedi-Heidari F, Marzban A, Raeisi-Ardali SR. Comparing the effect of emotional freedom technique on sleep quality and happiness of women undergoing breast cancer surgery in military and nonmilitary families: A quasi-experimental multicenter study. Perspect Psychiatr Care. 2022 Oct;58(4):2986-2997. doi: 10.1111/ppc.13150. Epub 2022 Oct 3. PMID 36192125
- [Background] Kang YS, Choi SY, Ryu E. The effectiveness of a stress coping program based on mindfulness meditation on the stress, anxiety, and depression experienced by nursing students in Korea. Nurse Educ Today. 2009 Jul;29(5):538-43. doi: 10.1016/j.nedt.2008.12.003. Epub 2009 Jan 13. PMID 19141364
- [Background] Kaur Khaira M, Raja Gopal RL, Mohamed Saini S, Md Isa Z. Interventional Strategies to Reduce Test Anxiety among Nursing Students: A Systematic Review. Int J Environ Res Public Health. 2023 Jan 10;20(2):1233. doi: 10.3390/ijerph20021233. PMID 36673999
- [Background] Lakens D. Calculating and reporting effect sizes to facilitate cumulative science: a practical primer for t-tests and ANOVAs. Front Psychol. 2013 Nov 26;4:863. doi: 10.3389/fpsyg.2013.00863. PMID 24324449
- [Background] Latifah, L., & Ramawati, D. (2018). Intervensi Emotional Freedom Technique (Eft) Untuk Mengurangi Nyeri Post Operasi Sectio Caesaria (Sc). Indonesian Nursing Journal Of Education And Clinic (INJEC), 1(1), 53-60.
- [Background] McCormick, S., & Lamberson, J. (2024). Interventions for test anxiety in nursing students: A literature review. Teaching and Learning in Nursing, 19(2), e404-e411.
- [Background] Menevse S, Yayla A. Effect of Emotional Freedom Technique Applied to Patients Before Laparoscopic Cholecystectomy on Surgical Fear and Anxiety: A Randomized Controlled Trial. J Perianesth Nurs. 2024 Feb;39(1):93-100. doi: 10.1016/j.jopan.2023.07.006. Epub 2023 Oct 6. PMID 37804271
- [Background] Moore-Hafter, B., Barbee, J., Zacharias-Miller, C., Shaner, L., & EFT International Executive, Research, Accreditation and Training Boards. (2023, November). Free tapping manual: A comprehensive introductory guide to EFT (Emotional Freedom Techniques) (Version 3.3.1). EFT International. https://eftinternational.org/what-is-eft-tapping
- [Background] Pandey, N. (2020). Eft As a Tool To Resolve Anxiety: a Case Study Approach. International Journal of PsychoSocial Research (IJPSR), 9(1).
- [Background] Patterson SL. The effect of emotional freedom technique on stress and anxiety in nursing students: A pilot study. Nurse Educ Today. 2016 May;40:104-10. doi: 10.1016/j.nedt.2016.02.003. Epub 2016 Feb 7. PMID 27125158
- [Background] Quinn BL, Peters A. Strategies to Reduce Nursing Student Test Anxiety: A Literature Review. J Nurs Educ. 2017 Mar 1;56(3):145-151. doi: 10.3928/01484834-20170222-05. PMID 28263352
- [Background] Rückert, H. W. (2015). Students׳ mental health and psychological counselling in Europe. Mental Health & Prevention, 3(1-2), 34-40.
- [Background] Salicru, S. (2025). Emotional freedom techniques in mental health care: evidence review, gaps, and future directions. Academia Mental Health and Well-Being, 2(2).
- [Background] Stapleton, P. (2019). The science behind tapping: A proven stress management technique for the mind and body. Hay House, Inc.
- [Background] Şahin, A. (2019). State test anxiety scale (STAS): Validity and reliability study. Trakya Eğitim Dergisi, 9(1), 78-90.
- [Background] Uzel, A., Emül, T. G., Yılmaz, D. V., Erdoğan, S., & Gürel, R. (2017). Determination of the effect of exam anxiety levels of the students the school nursing and midwifery on academic success Researcher, 5(4), 41-52.
- [Background] von der Embse N, Jester D, Roy D, Post J. Test anxiety effects, predictors, and correlates: A 30-year meta-analytic review. J Affect Disord. 2018 Feb;227:483-493. doi: 10.1016/j.jad.2017.11.048. Epub 2017 Nov 13. PMID 29156362
- [Background] Irmak Vural P, Aslan E. Emotional freedom techniques and breathing awareness to reduce childbirth fear: A randomized controlled study. Complement Ther Clin Pract. 2019 May;35:224-231. doi: 10.1016/j.ctcp.2019.02.011. Epub 2019 Feb 15. PMID 31003663
- [Background] Vural, P. I., Körpe, G., & Inangil, D. (2019). Emotional freedom techniques (EFT) to reduce exam anxiety in Turkish nursing students. European Journal of Integrative Medicine, 32, 101002.
- [Background] WMA (2013). Declaration of Helsinki "Ethical Principles for Medical Research Involving Human Subjects,"64th WMA General Assembly, Fortaleza, Brazil, in October 2013, https://www.wma.net/wp- content/uploads/2024/10/DoH-Oct2013.pdf
- [Background] Zheng D, Lin X, Gao X, Wang L, Zhu M. The impact of emotional freedom techniques on anxiety, depression, and anticipatory grief in people with cancer: A meta-analysis and systematic review. J Psychosom Res. 2025 May;192:112088. doi: 10.1016/j.jpsychores.2025.112088. Epub 2025 Mar 7. PMID 40073789